CLINICAL TRIAL: NCT02523963
Title: Effects of Family Work Shop for Children With Developmental Delays
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Ru-Lan Hsieh, Associate professor, Taipei Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H10427
Record Dates: First submitted 2015-08-07; First posted 2015-08-14 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-08

CONDITIONS: Developmental Delays
Keywords: family work shop

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- study group (Experimental): children with developmental delays participated 6 sessions of family work shop
  1. The family work shop has 5 courses, with 6 families in one course.
  2. Intervention of one course: 2-3 hours per session, one time per week, for a total of 6 weeks.
  Interventions: Other: family work shop
- control (No Intervention): children with normal development not participate the work shop followed up at before, and 6 weeks later

INTERVENTIONS:
Other: family work shop — 1. The family work shop has 5 courses, with 6 families in one course.
  2. One course of intervention: 2-3 hours per session, one time per week, for a total of 6 sessions in 6 week periods
  Arms: study group

SUMMARY:
The purpose of this study is to identify the effects of family work shop for children with developmental delays.

DETAILED DESCRIPTION:
Methods：

1. The family work shop has 5 courses, with 6 families in one course. 2. Intervention: 2-3 hours per session, one time per week, for a total of 6 weeks.

Effect：

1. Investigate the effects of family work shop for children with developmental delays, including health related quality of life, functional performance.
2. Investigate the effects of family care giver strain on family work shop for parents of children with developmental delays.
3. Investigate the differences of family impact between children with development delays and children with normal development.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of developmental delays and must be able to attend 6 weeks of work shop

Exclusion Criteria:

* Failed to obtain written informed consent

Ages: 18 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-01 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
change in health related quality of life questionnaire | baseline and 6 weeks
  to identify the changes of health related quality of life of children after the workshop

CONTACTS AND LOCATIONS:
Overall Officials: Ru-Lan Hsieh, MD, Principal Investigator — visiting staff of Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan